CLINICAL TRIAL: NCT06327269
Title: Innovative Diagnosis and Therapy in LDLT Patients With High-risk Hepatocellular Carcinoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MOHW111-TDU-B-221-114009
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: High Risk of Recurrence
Keywords: living donor liver transplantation (LDLT); hepatocellular carcinoma (HCC); PET; proton; yttrium 90; Lenvatinib; adjuvant treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A new generation of targeted therapies and adjuvant therapy after LDLT. (Active Comparator): The proton therapy or yttrium 90 as a more aggressive down-staging therapy may contribute to change tumor behavior. Lenvatinib is applied to adjuvant therapy after LDLT.
  Interventions: Drug: Lenvatinib 10 mg
- prolong the recurrence-free survival to high risk of HCC after LDLT (Active Comparator): Lenvatinib which is applied to adjuvant therapy after LDLT may prolong the recurrence-free survival
  Interventions: Drug: Lenvatinib 10 mg

INTERVENTIONS:
Drug: Lenvatinib 10 mg — Lenvatinib would be used on patients with advanced liver cancer after Liver transplantation as an adjuvant treatment.
  Other Names: Lenvima®

SUMMARY:
The challenge of LDLT to HCC is that tumors with a high risk of recurrence have a high rate of recurrence after liver transplantation, and there is no appropriate treatment to prevent HCC recurrence after transplantation in these patients. Using the advance proton therapy or yttrium 90 as a more aggressive down-staging therapy may contribute to change tumor behavior. It can be used to get a better treatment response and tumor necrosis before LDLT. As a result, it will improve recurrence-free survival and overall survival rate, especially in high-risk groups. In addition, lenvatinib is approved for using in patients with advanced liver cancer because its overall survival rate is not less than sorafenib in clinical trials. A new generation of targeted therapies will be applied to adjuvant therapy after LDLT.

ELIGIBILITY:
Inclusion Criteria

* Targeted therapy is acceptable within 1-2 months after liver transplantation.
* Immunosuppressive regimen consists of calcineurin inhibitor, mycophenolate mofetil and sirolimus.
* All male and female participants must take reliable contraceptive measures during the trial and within four weeks after the end of the trial.
* The definition of high-risk patients:
* The PET scan is positive before LDLT;
* Tumors beyond USCF criteria
* Poorly-differentiated tumor;
* The patients who has poor AFP response (<15%)or AFP>400 ng/ml after LRT after conventional LRT (RFA、PEI or TACE)

Exclusion Criteria

* Life expectancy is less than 3 months
* Patients are with other malignant tumors simultaneously.
* Patients are anaphylaxis to the inactive ingredients of lenvatinib or drugs.
* Pregnant or lactating women (Female participants need pregnancy test within 7 days before treatment).
* Preoperative history of severe cardiovascular disease: congestive heart failure > NYHA grade 2; active coronary heart disease (myocardial infarction occurred within 6 months before entry into the study); severe arrhythmia requiring antiarrhythmic treatment (allowable use of beta-blockers or digoxin); uncontrolled hypertension.
* History of HIV infection.
* Severe clinical active infections (> NCI-CTCAE version 3.0).
* Epilepsy patients requires medication (e.g. steroids or antiepileptic drugs).
* Patients with kidney diseases requires renal dialysis.
* Drug abuse, medical symptoms, mental illness or social status that may interfere with participants' participation in research or evaluation of research results.
* Patients who could not swallow oral drugs, such as those with severe upper gastrointestinal obstruction and need gastric tube feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival with adjuvant therapy | 2 years
  Lenvatinib treatment may prolong the recurrence-free survival rate after LDLT.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Kaohsiung City, Taiwan

REFERENCES:
- [Result] Han B, Ding H, Zhao S, Zhang Y, Wang J, Zhang Y, Gu J. Potential Role of Adjuvant Lenvatinib in Improving Disease-Free Survival for Patients With High-Risk Hepatitis B Virus-Related Hepatocellular Carcinoma Following Liver Transplantation: A Retrospective, Case Control Study. Front Oncol. 2020 Dec 7;10:562103. doi: 10.3389/fonc.2020.562103. eCollection 2020. PMID 33365268